CLINICAL TRIAL: NCT06514625
Title: Effect of Splinting and Kinesiotaping Treatments on Functional Status, Sleep Quality and Median Nerve Cross-sectional Area in Carpal Tunnel Syndrome: a Single Blind Prospective Randomized Controlled Study
Brief Title: Sleep Quality in Carpal Tunnel Syndrome, Splinting and Kinesiotaping
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konya Beyhekim Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 79735520-799
Record Dates: First submitted 2024-07-08; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Splints

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- splint and exercise (Experimental): The patient was asked to wear the fabricated splint that fixes the wrist in the neutral position every night and during the day as much as possible
  Interventions: Device: splint
- kinesiotaping and exercise (Experimental): Kinesiotaping was applied twice a week for a total of 8 sessions for 4 weeks. Taping was performed with a "neural technique" for the median and "field correction technique" for releasing the carpal tunnel. The elbow was positioned in full extension, the forearm in supination, and the wrist in 30 extension. I tape was used for neural technique. Tape was applied to the skin along the median nerve from the second and third metacarpophalangeal joints to five centimetres distal to the medial epicondyle. For the area correction technique, the I tape, which is half of the wrist circumference, was heavily stretched to the volar side of the wrist and the middle 1/3 part was taped without stretching the edges.
  Interventions: Device: splint
- exercise (Active Comparator): Nerve tendon gliding exercises were taught practically by an experienced physiotherapist. Participants were asked to do three sets of 10 repetitions every day for one month. Tendon gliding exercises were performed by bringing the hand into five different positions: regular grip, hook grip, punch, tabletop, and regular punch. Nerve gliding exercises were performed by bringing the fingers and wrist into six different positions: fingers and thumb in flexion with the wrist in neutral position, fingers and thumb in extension with the wrist in neutral position, thumb in neutral position with the wrist and fingers in extension, wrist, fingers, and thumb in extension, forearm in supination, and gentle stretching of the thumb with the other hand. Patients were given a thirty day exercise diary.
  Interventions: Device: splint

INTERVENTIONS:
Device: splint — ready night splints

SUMMARY:
The effect of conservative treatments on sleep quality in carpal tunnel syndrome is unclear.

Comparing the effect of splinting and kinesiotaping in carpal tunnel syndrome on functional status, pain, grip strength, nerve cross-sectional area and sleep quality.

Participants were divided into 3 groups. One group received night splint and nerve tendon gliding exercises, one group received kinesiotaping and nerve tendon gliding exercises, and one group received only nerve tendon gliding exercises. Participants were evaluated by a blinded investigator at baseline and at 3 months by Visual Analogue Scale (VAS), Boston Carpal Tunnel Syndrome Questionnaire, Pittsburgh Sleep Quality Index (PSQI), Jamar hand dynamometer and ultrasonography.

ELIGIBILITY:
Inclusion Criteria

* Being diagnosed with mild and moderate carpal tunnel syndrome with nerve conduction velocity study
* To be between the ages of 18-65

Exclusion Criteria:

* Inflammatory disease (rheumatoid arthritis, tendinitis, etc.),
* Osteoarthritis in the hand/wrist,
* Musculoskeletal conditions (hand, elbow, wrist),
* Thyroid disease
* Chronic kidney failure
* Carpal tunnel syndrome surgery,
* History of surgery and/or trauma to the upper extremity and neck.
* Pregnancy or diabetes-related carpal tunnel syndrome,
* Receiving any treatment for carpal tunnel syndrome (splint therapy, electrophysical agents, exercise, local corticosteroid injection) up to 3 months prior to the tests.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
sleep quality | at baseline and third month
  Evaluated with "The Pittsburgh Sleep Quality Index ".
median nerve cross-sectional area | at baseline and third month
  Measured at the wrist by ultrasonography.

CONTACTS AND LOCATIONS:
Locations (1):
- Konya Beyhekim Research and Training Hospital, Konya, Selçuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Karpuz S, Yilmaz R, Ozkan M, Kaya IC, Bulut O, Erol K, Yilmaz H. Effect of splinting and kinesiotaping treatments on functional status, sleep quality and median nerve cross-sectional area in carpal tunnel syndrome: A single blind prospective randomized controlled study. J Hand Ther. 2025 Jul-Sep;38(3):483-491. doi: 10.1016/j.jht.2024.12.001. Epub 2025 Jan 6. PMID 39765425